CLINICAL TRIAL: NCT01050855
Title: Reduced Intensity Conditioning (RIC) Regimen for Patients With Non-malignant Disorders
Acronym: RIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-005658; CHP 894 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Non Malignant Diseases; Immunodeficiencies; Hemoglobinopathies
Keywords: Non-malignant diseases; Immune deficiencies; Hemoglobinopathies; Reduced Intensity Conditioning(RIC)
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Hemoglobinopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- RIC: Distal Campath (Experimental): Day Treatment
  Day - 22 Inpatient: Alemtuzumab (Campath) test dose IV or SQ (subcutaneously) (subcutaneously) over 2 hours
  Day - 21 to-19 Alemtuzumab IV/ SQ (subcutaneously)
  Day - 7 to -3 Readmission to hospital Fludarabine IV
  Day - 2 Melphalan IV
  Day - 1 Begin cyclosporine infusion
  Day 0 Transplant: Bone marrow or cord blood infusion
  Interventions: Drug: RIC: Distal Campath
- RIC:Intermediate Campath (Experimental): Day Treatment
  Day - 14 to-10 Inpatient: Alemtuzumab (Campath) IV or SQ (subcutaneously)
  Day - 7 to -3 Fludarabine IV
  Day - 2 Melphalan 140 mg/m2 IV
  Day - 1 Cyclosporine infusion starts
  Day 0 Transplant: Bone marrow or cord blood infusion
  Interventions: Drug: RIC:Intermediate Campath
- RIC: Mini Busulfan (Experimental): Day Treatment
  Day - 8 Alemtuzumab (Campath) IV or SQ (subcutaneously)
  Day - 7 Alemtuzumab (Campath) IV or SQ (subcutaneously)
  Day - 6 Alemtuzumab (Campath) IV or SQ (subcutaneously) Busulfan IV Fludarabine IV
  Day - 5 Alemtuzumab (Campath) IV or SQ (subcutaneously) Busulfan IV Fludarabine IV
  Day - 4 Alemtuzumab (Campath) IV or SQ (subcutaneously) Fludarabine IV
  Day - 3 Fludarabine IV
  Day - 2 Fludarabine IV Cyclosporine infusion
  Day - 1 Rest
  Day 0 Transplant: Bone marrow or cord blood infusion
  Interventions: Drug: RIC: Mini Busulfan

INTERVENTIONS:
Drug: RIC: Distal Campath — Campath, Fludarabine, Melphalan, Cyclosporine, Cellcept (MMF)
  Other Names: Reduced Intensity Conditioning Regimen
  Arms: RIC: Distal Campath
Drug: RIC:Intermediate Campath — Campath, Fludarabine, Melphalan, Cyclosporine, Cellcept (MMF)
  Other Names: Reduced Intensity Conditioning Regimen
  Arms: RIC:Intermediate Campath
Drug: RIC: Mini Busulfan — Campath, Fludarabine, Busulfan, Cyclosporine, Cellcept (MMF)
  Other Names: Reduced Intensity Conditioning Regimen
  Arms: RIC: Mini Busulfan

SUMMARY:
This is a Phase II pilot study to evaluate engraftment and toxicity of patients with non-malignant diseases using a reduced intensity conditioning regimen in the setting of allogeneic transplant for non malignant diseases. Bone Marrow or cord blood will be acceptable as a stem cell source.

Recently, reduced intensity conditioning (RIC) regimens have been used for both adult patients with leukemias and pediatric patients with non-malignant diseases. These regimens are better tolerated, resulting in less transplant related morbidity and mortality. Stable mixed chimerism, while insufficient for eradication of leukemias, may be sufficient to cure patients with non-malignant diseases.

DETAILED DESCRIPTION:
There are two conditioning regimens in this protocol for children >6 months. Alemtuzumab (Campath), Fludarabine and Melphalan are used. The regimens differ by the timing and dosing of Alemtuzumab (Campath). The two timings are distal and intermediate.

* Distal campath is initiated 22 days prior to the allogeneic transplant.
* Intermediate campath is initiated 14 days prior to allogeneic transplant.

The conditioning regimen for children with immunodeficiencies <6 months omits melphalan, and substitutes two days of busulfan. This regimen is successfully used in the United Kingdom, and has been successful in a 3 month old infant at the Children's Hospital of Philadelphia (CHOP) who engrafted with a haploidentical donor.

ELIGIBILITY:
Inclusion Criteria:

1. Age >6 months- 25 years
2. Diseases eligible for Distal Alemtuzumab:

   * Immunodysregulation polyendocrinopathy enteropathy X-linked (IPEX) syndrome
   * Sickle cell disease
   * Thalassemia major
   * Bone marrow failure
3. Diseases eligible for Intermediate Alemtuzumab

   * Hemophagocytic lymphohistiocytosis other macrophage activation syndromes, severe Langerhans histiocytosis
   * Severe combined immune deficiency, adenosine deaminase deficiency, common variable immunodeficiency
   * Wiskott-Aldrich syndrome
4. Organ criteria:

   * Cardiac: Echocardiogram shortening fraction >27%
   * Renal: Serum creatinine less than 1.5 times the upper limit of normal for age
   * Hepatic: liver function tests must be less than 5 times the upper limit of normal
5. No active infections

Exclusion criteria

1. Uncontrolled bacterial, fungal or viral infections

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-01; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Engraftment | Post Transplant -100 days
  engraftment of patients with non-malignant disorders will be evaluated using a reduced-intensity conditioning regimen

SECONDARY OUTCOMES:
Survival | 1 year post transplant
  Event free survival will be evaluated by the time interval to either the primary or late graft failure, disease recurrence or death.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Olson, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] King AA, Kamani N, Bunin N, Sahdev I, Brochstein J, Hayashi RJ, Grimley M, Abraham A, Dioguardi J, Chan KW, Douglas D, Adams R, Andreansky M, Anderson E, Gilman A, Chaudhury S, Yu L, Dalal J, Hale G, Cuvelier G, Jain A, Krajewski J, Gillio A, Kasow KA, Delgado D, Hanson E, Murray L, Shenoy S. Successful matched sibling donor marrow transplantation following reduced intensity conditioning in children with hemoglobinopathies. Am J Hematol. 2015 Dec;90(12):1093-8. doi: 10.1002/ajh.24183. Epub 2015 Oct 6. PMID 26348869